CLINICAL TRIAL: NCT00005292
Title: Alpha1-antitrypsin Deficiency Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2014
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2004-08

CONDITIONS: Lung Diseases; Emphysema; Alpha-1 Antitrypsin Deficiency; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases; Emphysema; alpha 1-Antitrypsin Deficiency; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To collect data from the 37 participating clinical centers on patients with alpha1-antitrypsin deficiency, including those who received replacement therapy with an intravenous preparation of alpha1-proteinase inhibitor (A1Pi) concentrate.

DETAILED DESCRIPTION:
BACKGROUND:

Severe congenital deficiency for alpha1-antitrypsin is associated with the early onset of emphysema, usually by the third decade of life. One approach to correct this deficiency is though replacement with alpha1-antitrypsin (referred to as alpha1-proteinase (A1Pi) inhibitor in its purified form). An intravenous preparation of A1Pi concentrate was produced from human plasma by Cutter Biological, a division of Miles, Inc., Berkeley, California. This preparation had been evaluated in a clinical study for its safety and biochemical efficacy. Based on the augmentation of its levels in the lung upon intravenous administration, the A1Pi preparation was licensed by the Food and Drug Administration for replacement therapy to treat individuals with severe congenital deficiency and impaired lung function. When the registry began in 1988, clinical efficacy was plausible, but unproven and there was no data base for estimating the degree of clinical benefit, if any.

Slow progression of emphysema and lack of an adequate control group have made it difficult to evaluate the proteinase inhibitor through a controlled clinical trial. A patient registry was an alternative method to collect data on the effect of long-term replacement therapy with A1Pi on rate of decline of lung function. The registry also included individuals who did not receive the replacement therapy in order to obtain a better knowledge of the rate of decline of lung function associated with the congenital deficiency for alpha1-antitrypsin.

DESIGN NARRATIVE:

The registry consisted of a clinical coordinating center, 37 participating clinical centers that contributed patient data to the registry, a steering committee, and a data analysis and policy board, both appointed by the National Heart, Lung, and Blood Institute. Data collected on all patients included a clinical history, laboratory evaluations such as chest x-ray, lung function studies of vital capacity, total lung capacity, forced expiratory volume in one second (FEV1) and blood studies. In addition, patients receiving replacement therapy had baseline lung function tests, spirometry every six months following initiation of replacement therapy, and measurements of serum alpha1-antitrypsin level pre- and post-infusion, once every six months. The recruitment phase ended in September 1990. Support for the registry ended in June, 1998.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-09; Study Completion 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schluchter — The Cleveland Clinic

REFERENCES:
- [Background] Stoller JK, Williams GW, Crystal RG. Alpha 1-antitrypsin deficiency registry. Chest. 1990 May;97(5):1278. doi: 10.1378/chest.97.5.1278b. No abstract available. PMID 2331946
- [Background] Schluchter MD. Methods for the analysis of informatively censored longitudinal data. Stat Med. 1992 Oct-Nov;11(14-15):1861-70. doi: 10.1002/sim.4780111408. PMID 1480878
- [Background] A registry of patients with severe deficiency of alpha 1-antitrypsin. Design and methods. The Alpha 1-Antitrypsin Deficiency Registry Study Group. Chest. 1994 Oct;106(4):1223-32. PMID 7924498
- [Background] Stoller JK, Buist AS, Burrows B, Crystal RG, Fallat RJ, McCarthy K, Schluchter MD, Soskel NT, Zhang R. Quality control of spirometry testing in the registry for patients with severe alpha1-antitrypsin deficiency. alpha1-Antitrypsin Deficiency Registry Study Group. Chest. 1997 Apr;111(4):899-909. doi: 10.1378/chest.111.4.899. PMID 9106567
- [Background] McElvaney NG, Stoller JK, Buist AS, Prakash UB, Brantly ML, Schluchter MD, Crystal RD. Baseline characteristics of enrollees in the National Heart, Lung and Blood Institute Registry of alpha 1-antitrypsin deficiency. Alpha 1-Antitrypsin Deficiency Registry Study Group. Chest. 1997 Feb;111(2):394-403. doi: 10.1378/chest.111.2.394. PMID 9041988
- [Background] Turino GM, Barker AF, Brantly ML, Cohen AB, Connelly RP, Crystal RG, Eden E, Schluchter MD, Stoller JK. Clinical features of individuals with PI*SZ phenotype of alpha 1-antitrypsin deficiency. alpha 1-Antitrypsin Deficiency Registry Study Group. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 1):1718-25. doi: 10.1164/ajrccm.154.6.8970361.
- [Background] Schluchter MD, Stoller JK, Barker AF, Buist AS, Crystal RG, Donohue JF, Fallat RJ, Turino GM, Vreim CE, Wu MC. Feasibility of a clinical trial of augmentation therapy for alpha(1)-antitrypsin deficiency. The Alpha 1-Antitrypsin Deficiency Registry Study Group. Am J Respir Crit Care Med. 2000 Mar;161(3 Pt 1):796-801. doi: 10.1164/ajrccm.161.3.9906011. PMID 10712324
- [Background] Survival and FEV1 decline in individuals with severe deficiency of alpha1-antitrypsin. The Alpha-1-Antitrypsin Deficiency Registry Study Group. Am J Respir Crit Care Med. 1998 Jul;158(1):49-59. doi: 10.1164/ajrccm.158.1.9712017. PMID 9655706
- [Background] Eden E, Hammel J, Rouhani FN, Brantly ML, Barker AF, Buist AS, Fallat RJ, Stoller JK, Crystal RG, Turino GM. Asthma features in severe alpha1-antitrypsin deficiency: experience of the National Heart, Lung, and Blood Institute Registry. Chest. 2003 Mar;123(3):765-71. doi: 10.1378/chest.123.3.765. PMID 12628876
- Available data/document: Individual Participant Data Set: AADR — http://biolincc.nhlbi.nih.gov/studies/aadr — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — https://biolincc.nhlbi.nih.gov/studies/aadr/Forms/